CLINICAL TRIAL: NCT02491671
Title: Prospective, Multicenter, Open-Label, Randomized, Phase III Clinical Trial of Prevention of Prolonged Air Leak After Lung Resection in High-risk Patients, Applying HEMOPATCH®
Brief Title: Effectiveness Novel Tissue Sealant, Prevention Prolonged Air Leak (PAL) After Lung Resection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other)
Collaborators: Instituto de Investigación Biomédica de Salamanca (Other); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HEMOPATCH/FAP/2014
Record Dates: First submitted 2015-06-10; First posted 2015-07-08 (Estimated); Results first posted 2021-07-27 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Prolonged Air Leak; Lung Resection
Keywords: Prevention PAL Prolonged Air Leak (PAL); Lung Resection; Thoracic Surgery; Post-operative Thoracic Air Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Experimental group: At the end of lung resection, lung sutures and 1.5 cm of lung parenchyma on each side will be covered by Hemopatch. No additional measures for preventing air leak will be indicated. In the case of massive air leak in spite of the use of Hemopatch, each surgeon will decide on the indication of additional sutures of tissue plasties. These cases will be accounted for failures on an intention to treat basis.
  Interventions: Device: Hemopatch; Procedure: standard preventive measures
- Control group (Other): Control group: The standard preventive measures will be followed in each center, including reinforcement of sutures, pleural tents, suturing pericardial or subcutaneous fat
  Interventions: Procedure: standard preventive measures

INTERVENTIONS:
Device: Hemopatch
  Arms: Experimental group
Procedure: standard preventive measures

SUMMARY:
The effectiveness of tissue sealants to prevent Prolonged Air Leak (PAL) after lung resection procedures remains unproved. The investigators hypothesize that one of the main reasons for that is the heterogeneity of previously studied populations. Since currently the risk of postoperative PAL can be scored with a reasonable accuracy, the aim of this research is to investigate the effect of routine application of a novel tissue sealant in patients selected on the basis of a high risk of PAL estimated before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled anatomical lung resection indicated for any non-infectious disease (excluding Pneumonectomy)
* Patients classified in class D according estimated risk of PAL
* Age between 18 and 80 years

Exclusion Criteria:

* Those patients that according to Investigator assessment are not going to tolerate the procedure
* Clinical and anesthetic criteria that contraindicate surgery
* Severe uncontrolled illness
* Pregnancy
* Patients that are under Investigational New Drug treatment or have participated in study with a investigational drug (authorized or not) in 30 days before randomization.
* Lack of Informed Consent or patient refusal
* Postsurgery mechanical ventilation or repeated surgery in follow-up month.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Varela, MD PhD FETCS, Study Director — IBSAL-Instituto de Investigación Biomédica de Salamanca
Locations (6):
- Spain (6):
  - Hospital Universitario Marqués de Valdecilla de Santander, Santander, Cantabria
  - Hospital Clinic, Barcelona
  - Hospital Universitario Ramón y Cajal de Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario de Salamanca (CAUSA), Salamanca
  - Hospital Universitario Virgen del Rocío, Seville

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Group: Experimental group: At the end of lung resection, lung sutures and 1.5 cm of lung parenchyma on each side will be covered by Hemopatch. No additional measures for preventing air leak will be indicated. In the case of massive air leak in spite of the use of Hemopatch, each surgeon will decide on the indication of additional sutures of tissue plasties. These cases will be accounted for failures on an intention to treat basis.
  Hemopatch
  standard preventive measures
- Control Group: Control group: The standard preventive measures will be followed in each center, including reinforcement of sutures, pleural tents, suturing pericardial or subcutaneous fat
  standard preventive measures
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 129 | 131
Completed | 118 | 118
Not Completed | 11 | 13
Not completed — Adverse Event | 6 | 8
Not completed — Death | 0 | 2
Not completed — Use of sealants other than Hemopatch | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 118 | 118 | 236
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 70.77 [52.26 to 83.63] | 70.76 [49.21 to 83.41] | 70.77 [51 to 83.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 52
  Male | 93 | 91 | 184
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Spain | 118 | 118 | 236
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 24.5 [18 to 34] | 24.27 [17.47 to 39.8] | 24.4 [17.5 to 37]
American Society of Anesthesiologists (ASA) classification [Count of Participants; unit: Participants] — ASA 2: A moderate but definite systemic disturbance.
  ASA 3: Severe systemic disturbance from any cause or causes. It is not possible to state an absolute measure of severity, as this is a matter of clinical judgment.
  ASA 4: Extreme systemic disorders which have already become an eminent threat to life regardless of the type of treatment. Because of their duration or nature there has already been damage to the organism that is irreversible. This class is intended to include only patients that are in an extremely poor physical state.
  Participants
    ASA 2 | 54 | 51 | 105
    ASA 3 | 62 | 65 | 127
    ASA 4 | 2 | 2 | 4
Type of Surgery [Count of Participants; unit: Participants]
  Segmentectomy | 7 | 4 | 11
  Lobectomy | 106 | 107 | 213
  Bilobectomy | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Prolonged Air Leak (PAL)
Description: Prevalence of Prolonged Air Leak (PAL) measured as binary variable (YES/NO) and recorded, from day of surgery to the fifth postoperative day, in the study questionnaire. The occurrence of the outcome will be recorded if air leak exists 5 days or more after surgery
Time Frame: From day of surgery to the fifth postoperative day
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 118 | 118
Participants | 33 | 24
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Superiority; p = 0.171, Chi-squared; Risk Ratio (RR) = 1.219, 95% CI 2-sided [0.891 to 1.583]

2. Secondary Outcome: Duration of Air Leaks
Description: Measured as continuous variable (days) and recorded, from day of surgery to the day of withdraw the chest tube. (standardized criteria for pulling out chest drainage/s will be agreed among investigators)
Time Frame: Check everyday from day of surgery up to 38 days post-operative at maximum
Measure: Mean (Full Range); unit: days
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 118 | 118
days | 1 [0 to 12] | 1 [0 to 38]
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Superiority; p > 0.05, Wilcoxon (Mann-Whitney); z = 0.288 — Wilcoxon rank-sum (Mann-Whitney) test Unadjusted variance 274999.00 Adjustment for ties --21069.78 Adjusted variance 253929.22 z = 0.288; Prob > |z| = 0.7735

3. Secondary Outcome: Number of Participants With at Least One Chest Tube Reinsertion
Description: Rate of patients needing postoperative reinsertion of chest drainages due to symptomatic pneumothorax. Following daily during hospital stay and pone follow-up until 30th day post-operative.
Time Frame: From day of surgery up to 30 days thereafter
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 118 | 118
Participants | 3 | 6
Statistical Analysis 1: Comparison: Experimental Group vs Control Group; Test type: Superiority; p = 0 .307, Chi-squared; Risk Ratio (RR) = 1.351, 95% CI 2-sided [0.657 to 1.879]

4. Secondary Outcome: Number of Participants With One or More Readmission
Description: Rate of readmissions due to relapsing pneumothorax (follow-up 30 days)
Time Frame: 30 days post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 118 | 118
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Through study completion, a total of up to 3 months.
Arm/Group | Experimental Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/118 | 2/118
Serious Adverse Events (participants affected / at risk) | 3/118 | 7/118
Other Adverse Events (participants affected / at risk) | 0/118 | 0/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group (N=118) | Control Group (N=118)
Pulmonary. Mechanical ventilation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Reoperation for bleeding (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
Only the population in which a very high rate of PAL is expected was enrolled. There was no stratification by lung function or type of lung resection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-17): https://cdn.clinicaltrials.gov/large-docs/71/NCT02491671/Prot_SAP_000.pdf
  • Informed Consent Form (2015-03-03): https://cdn.clinicaltrials.gov/large-docs/71/NCT02491671/ICF_001.pdf